CLINICAL TRIAL: NCT01649492
Title: In Vivo Inhibition Profile of CYP2C9 by Pineapple Juice
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Isabelle Spriet, PharmD, PhD, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: S54465
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Healthy Volunteers
Keywords: diclofenac; CYP2C9; bromelain; pineapple juice

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- diclofenac without pineapple juice (No Intervention): single dose of diclofenac 25 mg without pre-exposure to pineapple juice
- diclofenac with pineapple juice (Active Comparator): single dose of diclofenac 25 mg with pre-exposure to pineapple juice
  Interventions: Dietary Supplement: pineapple juice (Carrefour n°1) 500 ml/day 5 days

INTERVENTIONS:
Dietary Supplement: pineapple juice (Carrefour n°1) 500 ml/day 5 days
  Arms: diclofenac with pineapple juice

SUMMARY:
The goal of this study is to evaluate the actual potential for in vivo pineapple juice inhibition with CYP2C9 substrates in human volunteers with use of diclofenac as a marker of CYP2C9 activity.

DETAILED DESCRIPTION:
For ovarian cancer, colorectal and gastric cancers presenting with peritoneal metastases, complete tumor removal at surgery is the most important independent prognostic factor. Consequently, accurate detection of tumors often compromising resectability, like extra-abdominal metastases, liver metastases, portal and superior mesenteric artery deposits and extensive intestinal serosal invasion is pivotal prior to treatment selection. Computed tomography (CT) has variable accuracy for staging, due to the difficult detection of low-contrast or small-sized peritoneal or nodal metastases. Fluorodeoxyglucose positron emission tomography/CT (FDG-PET/CT) improves detection of thoraco-abdominal lymphadenopathy and liver metastases, but inconsistently detects small (<5mm) peritoneal metastases. Therefore a diagnostic staging laparoscopy under general anesthesia is currently the necessary standard of clinical practice in addition to imaging for assessment of operability.

Whole body diffusion-weighted magnetic resonance imaging is researched at the department of radiology, University Hospitals Leuven in collaboration with the departments of abdominal surgery, oncologic surgery, oncologic gynaecology and digestive oncology. The technique holds high promise to combine a high accuracy in systemic thoraco-abdominal staging and peritoneal assessment of operability. Technological progress has enabled time-efficient WB-DWI with thin-slice-acquisition and multiplanar image reformatting. DWI depicts lesions by measuring water diffusion differences, correlating with cellular density. Tumors are depicted with high signal compared to background by combining a short-T1-inversion-time inversion recovery (STIR) prepulse - suppressing ascites, blood vessels, fat, bowel and visceral organs - and heavy diffusion weighting. However, due to contraction and mucosal cellularity, the bowel wall can show increased signal-intensity (SI), hampering the detection of serosal deposits. This is overcome by suppressing contractions by intravenous antispasmodic and by distending the bowel wall and suppressing the signal of bowel content by peroral pineapple juice which shows negative contrast properties due to the manganese-content. In a first pilot study in ovarian cancer at this center in 32 patients, an accuracy for detection of intestinal serosal metastases of 90% was reached by WB-DWI combined with peroral pineapple juice. As such, the pineapple juice plays a pivotal role as a peroral contrast in addition to WB-DWI for accurate peritoneal staging.

To date, the inhibitory potential of pineapple juice on cytochrome P450 2C9 activity has only been described in vitro in human microsomes. In this model, in which diclofenac and its metabolite 4-OH-diclofenac have been used as probes for CYP2C9 activity, it has been shown that pineapple juice is capable to inhibit CYP2C9 very potently (IC50 0.08%) in an irreversible manner. It has been suggested that the main effect is caused by bromelain, a 24-26 kDa cysteine protease enzyme present in pineapple juice. The intestinal absorption of intact bromelain after oral intake has been described in 19 healthy men, which is surprising as the adult intestinal epithelium has traditionally been described as non-permeable to proteins. The (limited) absorption is thought to occur via the paracellular route, which could explain that the catalytic activity bromelain is preserved following absorption into the blood circulation. Although no effects of bromelain on CYP2C9 activity are expected in vivo (due to low oral bioavailability), no in vivo trials have been undertaken to elucidate if pineapple juice, and more specifically bromelain, is capable of inhibiting intestinal and, more importantly, hepatic CYP2C9 in a clinically relevant manner.

The in vivo inhibitory profile of CYP2C9 by pineapple juice will be evaluated in this study in 10 healthy volunteers, by examining the impact on the area-under-the-curves (AUCs) of diclofenac and its metabolite 4-OH diclofenac.

ELIGIBILITY:
Inclusion Criteria:

* adult healthy volunteers

Exclusion Criteria:

* younger than 18 yrs
* older than 60 yrs
* pregnant or lactating women
* medical history of gastric or duodenal ulcers, gastro-oesofageal reflux disease, dyspepsia, asthma, any allergy to NSAIDS
* patients taking co-medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
a) AUC 4-OH-diclofenac / AUC diclofenac quantified in plasma, on days 1 (without pineapple juice) and 11 (after pretreatment with pineapple juice) | day 1 and day 11
  see above

SECONDARY OUTCOMES:
(b) AUC 4-OH-diclofenac/ AUC diclofenac quantified in urine, on days 1 (without pineapple juice) and 11 (after pretreatment with pineapple juice) | day 1 and day 11
  see above

OTHER OUTCOMES:
c) Bromelain activity quantified in plasma, measured on days 1 and 11 | day 1 and day 11
  see above

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PharmD PhD, Principal Investigator — Pharmacy Dpt, University Hospitals Leuven; Hans Prenen, MD PhD, Study Chair — Digestive Oncology, University Hospitals Leuven; Vincent Vandecaveye, MD PhD, Study Chair — Radiology Dpt, University Hospitals Leuven; Pieter Annaert, PharmD PhD, Study Chair — Laboratory for Pharmacotechnology and Biopharmacy, Catholic University Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium